CLINICAL TRIAL: NCT06994767
Title: Speech-derived Digital Biomarkers for Assessing Mild Cognitive Impairment and Alzheimer's Disease Diagnosis Accuracy
Brief Title: Speech-derived Digital Biomarkers Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Canary Speech Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2024-0418
Record Dates: First submitted 2025-05-13; First posted 2025-05-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment (MCI); Alzheimer Disease
Keywords: Vocal biomarkers; Mild Cognitive Impairment; Alzheimer's Disease; Deep machine learning; Artificial Intelligence application
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Validation Studies as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild Cognitive Impairment (MCI) (Experimental): Patients with a mild congitive impairment
  Interventions: Other: The Canary Application
- Alzheimer's Disease (Experimental): Patients with an Alzheimer's Disease diagnosis
  Interventions: Other: The Canary Application
- Healthy Volunteers (Active Comparator): Patients without a diagnosis of MCI or Alzheimer's, or other types of dementia
  Interventions: Other: The Canary Application

INTERVENTIONS:
Other: The Canary Application — The CANARY application will use clinically validated survey instruments and voice recordings to measure user MCI status /Alzheimer's data. These tests are designed to evaluate a user's voice characteristics and potentially identify disease-specific patterns.
  Other Names: Validation

SUMMARY:
The goal is to assess the accuracy of an application that analyzes voice characteristics to diagnose patients with mild cognitive impairment (MCI) and Alzheimer's disease (AD). The main question is whether the application's diagnosis is the same as the clinician's for MCI and AD patients.

DETAILED DESCRIPTION:
The study aims to assess the sensitivity and specificity of an application that uses vocal biomarkers to diagnose patients with mild cognitive impairment (MCI) and Alzheimer's disease. The application will use clinically validated survey instruments and voice recordings to determine the disease status of patients with MCI and Alzheimer's disease. The diagnosis developed by the application is the primary outcome variable. To determine the sensitivity and specificity, the application diagnosis will be compared against the physician's clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 50 and above
* Willing and capable of participating in all aspects of the study
* Willing and capable of giving informed consent
* Diagnosis of MCI or Alzheimer's by the physician
* For the control group: Without diagnosis of MCI or Alzheimer's or other types of dementia
* Subjects are free of any medical condition(s) that, according to exclusion criteria, might audibly affect voice characteristics
* Subject must be able to speak and read with fluency in the English language.

Exclusion Criteria:

* All participants below 50 years
* Failure to provide informed consent
* Individuals with the following medical conditions will be excluded:

  i) Parkinson's disease ii) Huntington's disease iii) Cancer and active cancer treatments
* Persons with speech characteristics (heavy accents, slurring, stuttering, etc.) that would interfere with voice recording or voice analysis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to assess the sensitivity biomarkers in patients with MCI and AD diagnosis | Upon enrollment
  The CANARY application will use clinically validated survey instruments and voice recordings to analyze the data and determine the patient's MCI/ Alzheimer's disease diagnosis. The diagnosis developed by the application is the primary outcome variable. To determine the sensitivity, the application diagnosis will be compared against the clinical diagnosis of the physician.
The primary objective of the study is to assess the specificity of vocal biomarkers in patients with MCI and AD diagnosis | Upon enrollment
  The CANARY application will use clinically validated survey instruments and voice recordings to analyze the data and determine the patient's MCI/ Alzheimer's disease diagnosis. The diagnosis developed by the application is the primary outcome variable. To determine the specificity, the application diagnosis will be compared against the clinical diagnosis of the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Sakshi Jain, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Sanchez F, Meilan JJG, Carro J, Ivanova O. A Prototype for the Voice Analysis Diagnosis of Alzheimer's Disease. J Alzheimers Dis. 2018;64(2):473-481. doi: 10.3233/JAD-180037. PMID 29914025
- [Background] Mueller KD, Hermann B, Mecollari J, Turkstra LS. Connected speech and language in mild cognitive impairment and Alzheimer's disease: A review of picture description tasks. J Clin Exp Neuropsychol. 2018 Nov;40(9):917-939. doi: 10.1080/13803395.2018.1446513. Epub 2018 Apr 19. PMID 29669461
- [Background] Garcia AM, de Leon J, Tee BL, Blasi DE, Gorno-Tempini ML. Speech and language markers of neurodegeneration: a call for global equity. Brain. 2023 Dec 1;146(12):4870-4879. doi: 10.1093/brain/awad253. PMID 37497623
- [Background] Sanborn V, Ostrand R, Ciesla J, Gunstad J. Automated assessment of speech production and prediction of MCI in older adults. Appl Neuropsychol Adult. 2022 Sep-Oct;29(5):1250-1257. doi: 10.1080/23279095.2020.1864733. Epub 2020 Dec 30. PMID 33377800
- [Background] Vinod Subramanian, Namhee Kwon, Raymond Brueckner, Nate Blaylock, Henry O'Connell,